CLINICAL TRIAL: NCT06032663
Title: Use of PET-MR in Head and Neck Cancer Patients - Diagnostic and Therapeutic Applications
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STH21185; 286722 (Other: IRAS)
Record Dates: First submitted 2023-09-04; First posted 2023-09-13 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Head and Neck Cancer
Keywords: Head; Neck; Cancer; PET MRI
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET-MRI within 1 week of planning scan. (Experimental): Patients would not normally have a PET-MRI as well as planning scan. In this experimental arm, patients will be given a PET-MRI within 1 week of the planning scan.
  Interventions: Diagnostic Test: PET-MRI

INTERVENTIONS:
Diagnostic Test: PET-MRI — Patients that participate in the current study will have an extra PET-MRI scan, which will expose them to a small amount (4 - 6 mSv) of extra radiation.

SUMMARY:
The primary research question to be answered in this project is "Are patients with locally-advanced head and neck cancer able to tolerate a PET-MRI scan when they are immobilised in a radiotherapy treatment shell?" This will be assessed by measuring the proportion of patients that complete the full scanning protocol and by obtaining participant feedback on their experience of completing the scan.

The secondary question is "Can a PET-MRI scan fused with a planning CT scan improve the accuracy in radiotherapy planning of patients with head and neck cancer? Accuracy will be assessed by:

1. Comparing the radiotherapy target volumes and radiotherapy plans with and without the use of a PET-MRI scan.
2. Comparing inter- and intra-observer variability in treatment contours with and without the use of a PET-MRI scan within and between oncologists and implications of that.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or over
2. Able to give informed written consent.
3. New diagnosis of biopsy-proven head and neck cancer.
4. WHO performance status ≤ 2.
5. MDT-recommended treatment with radical radiotherapy, with or without concurrent systemic therapy.
6. MRI and PET-CT staging scans for diagnosis.

Exclusion Criteria:

1. Known intolerance/sensitivity to 18F-2-deoxyglucose or gadolinium-containing contrast agents.
2. Claustrophobia or other contraindications to MRI.
3. Unable to pass through a 55 cm hula hoop.
4. Female patients that are pregnant or breastfeeding.
5. Unable to understand written or spoken English.
6. Patients not undergoing radical intent radiotherapy.
7. Patients with stage 4 or 5 chronic kidney disease or other biochemical abnormalities e.g. uncontrolled blood glucose levels which can have an impact on PET-MRI imaging or contrast administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Completion of PET-MRI | 12 months
  To assess the proportion of patients completing the full PET-MRI scans when they are immobilised in a radiotherapy treatment shell.

SECONDARY OUTCOMES:
Impact of additional PET-MRI on radiotherapy target volumes | 12 months
  The secondary objective is to compare the radiotherapy target volumes between conditions (with vs without the use of PET-MRI scan)
Impact of additional PET-MRI on treatment plan | 12 months
  Assess inter- and intra-observer variability in treatment contours and precision of target delineation in the three categories above (CT, CT-MRI, and CT-PET-MRI scans). This will be assessed using Hausdorff distance in the three categories.
Impact of additional PET-MRI on treatment plan | 12 months
  Assess inter- and intra-observer variability in treatment contours and precision of target delineation in the three categories above (CT, CT-MRI, and CT-PET-MRI scans). This will be assessed using Dice Similarity Index in the three categories.

OTHER OUTCOMES:
Added benefit to diagnostic investigations | 12 months
  Clinical reports of the PET-MRI scan will be compared to reports from staging MRI and PET-CT scans to determine if any new diagnostic information is brought to light by PET-MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Satya Garikipati, MD, Principal Investigator — STH Contracted Consultant
Locations (1):
- Cancer Research Centre at Weston Park Hospital, Sheffield, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD will not be available/shared outside the study

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/63/NCT06032663/Prot_SAP_000.pdf